CLINICAL TRIAL: NCT02274610
Title: Phase I Trial to Compare Pharmacokinetics and Safety of Docetaxel PNP With Taxotere in Subjects With Advanced Solid Tumor
Brief Title: Pharmacokinetic Study of Docetaxel-PNP and Taxotere to Treat Patient With Advanced Solid Cancer
Acronym: DOPNP201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DOPNP201
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2014-10

CONDITIONS: Solid Tumor
Keywords: docetaxel; Pharmacokinetic
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Period 1: Docetaxel-PNP / Washout: 3 weeks / Period 2: Taxotere
  Interventions: Drug: Docetaxel-PNP; Drug: Taxotere
- Group B (Experimental): Period 1: Taxotere / Washout: 3 weeks / Period 2: Docetaxel-PNP
  Interventions: Drug: Docetaxel-PNP; Drug: Taxotere

INTERVENTIONS:
Drug: Docetaxel-PNP — Docetaxel Polymeric Nanoparticle Formulation
Drug: Taxotere — Docetaxel

SUMMARY:
Evaluation of the pharmacokinetic equivalence of two Docetaxel formulations in terms of AUC and Cmax

DETAILED DESCRIPTION:
Comparison of pharmacokinetic parameters (T1/2β, CL, Vdss) Safety as measured by adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patient ages more than 18 years old
* Patient should voluntarily sign a written informed consent before study entry
* Patient historically or cytologically confirmed diagnosis of advanced solid tumor and patient with measurable disease or evaluable disease by RECIST criteria
* Progressive disease with development of new lesions or an increase in preexisting lesions or standard therapy in order to provide clinical benefit does not exist or is no longer effective
* Previous anti-cancer therapies must be completed before 21days of first study dose and Patient must have recovered from any previous therapy
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Patient has a life expectancy of at least 3 months
* Baseline studies for determining eligibility must be completed within 14 days of first study dose and patient has a adequate organ function including the following:

  * Hb ≥ 10g/dl
  * ANC ≥ 1.5 X 109/L
  * Platelet count ≥ 100 X 109/L
  * Serum total bilirubin ≤ 1.5 mg/dL
  * Serum AST and ALT ≤ 2.5 X UNL
  * Serum ALP ≤ 2.5ⅹUNL
  * Serum creatinine ≤ 1.5 X UNL

Exclusion Criteria:

* Patient has had a major surgery except tumor ablation within 2 weeks before screening visit
* Patient has a brain metastasis with neurologic symptom
* Patient has a sensory neuropathy or motor neuropathy ≥ grade 2 by NCI-CTCAE
* Patient has any serious concurrent disease such as:

Any medical or psychiatric condition that, in the opinion of the investigator, would prohibit the understanding and giving of informed consent Severe cardiovascular disease (e.g. ischemic heart disease requiring medication or myocardial infraction within the past six months, grade 3-4 congestive heart failure defined by the New York Heart Association criteria) Active un controlled infection.

* Patient has hypersensitivity to the Investigational product or their excipients
* Patient has participated in any other clinical trial within 4 weeks before screening visit
* Woman is pregnant or breast feeding
* Subjects who are of childbearing potential who do not use a medically acceptable method of birth control or do not agree to continue use of this method throughout the trial (screening, treatment period, and 3 weeks from the last done). A negative pregnancy test (urine or serum) should be documented within 14 days prior to initiation of trial medication for women of childbearing potential who have not been amenorrheic for at least 12 months prior to registration into the trial or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy). Medically acceptable methods include:

  * Barrier method with spermicide
  * Intrauterine device
  * Complete abstinence, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of DocetaxelPNP and Taxotere in terms of Area Under the Curve (AUC) | 3 months

SECONDARY OUTCOMES:
Elimination Half Life (T1/2) of DocetaxelPNP and Taxotere | 3 months
Clearance (CL) of DocetaxelPNP and Taxotere | 3 months
Volume of Distribution at steady state (Vdss) of DocetaxelPNP and Taxotere | 3 months
Number of participants with Adverse Events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mi-ryung Jin, Masters, Study Director — Samyang Biopharmaceuticals Corporation